CLINICAL TRIAL: NCT01242917
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of CCX354-C in Subjects With Rheumatoid Arthritis Partially Responsive to Methotrexate Therapy
Brief Title: A Study to Evaluate the Safety and Efficacy of CCX354-C in Subjects With Rheumatoid Arthritis Partially Responsive to Methotrexate Therapy
Acronym: CARAT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL004_354; 2010-019964-36 (EudraCT Number)
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CCX354-C 100mg twice daily (Experimental)
  Interventions: Drug: CCX354-C
- CCX354-C 200mg once daily (Experimental)
  Interventions: Drug: CCX-354-C

INTERVENTIONS:
Drug: CCX-354-C — 200mg film-coated tablets once daily for 12 weeks + Methotrexate
  Arms: CCX354-C 200mg once daily
Drug: Placebo — Placebo film-coated tablets twice daily for 12 weeks + methotrexate
  Arms: Placebo
Drug: CCX354-C — 100mg film-coated tablets twice daily for 12 weeks + methotrexate
  Arms: CCX354-C 100mg twice daily

SUMMARY:
This is a randomized, double-blind, placebo-controlled, Phase 2 study to evaluate the safety and efficacy of CCX354-C in subjects with rheumatoid arthritis partially responsive to methotrexate therapy.

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18-75 years inclusive, with functional class I to III rheumatoid arthritis (RA) based on American College of Rheumatology (ACR) criteria for at least 3 months prior to screening; wheel-chair bound subjects or those with irreversible disease will not be eligible;
2. Subjects must have active RA, defined by a minimum of 8 swollen joints and 8 tender/painful joints (based on 66/68 joint count), at screening
3. Serum C-reactive protein (CRP) above 5 mg/L at screening;
4. Must have been on methotrexate (7.5 to 25 mg/week) taken orally, subcutaneously, or intramuscularly for ≥ 16 weeks and on a stable dose for ≥ 8 weeks prior to randomization;
5. If on hydroxychloroquine, must have been on a stable dose for ≥ 16 weeks prior to randomization;
6. If taking non-steroidal anti-inflammatory drugs (NSAIDs), must have been on stable doses for ≥ 2 weeks before randomization;
7. If taking oral corticosteroids, subjects may not take more than 10 mg/day of prednisone or equivalent, and must have been on a stable dose for ≥ 4 weeks before randomization;
8. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
9. Negative result of the human immunodeficiency virus (HIV) screen, the hepatitis B screen, and the hepatitis C screen;
10. Judged to be otherwise healthy by the Investigator, based on medical history, physical examination (including electrocardiogram [ECG]), and clinical laboratory assessments;
11. Female subjects of childbearing potential, and male subjects with partners of childbearing potential, may participate if adequate contraception is used during, and for at least the four weeks after administration of study medication

Exclusion Criteria:

1. Diagnosed with RA prior to 16 years of age;
2. Women who are pregnant, breastfeeding, or have a positive serum pregnancy test at screening;
3. History within one year prior to randomization of illicit drug use;
4. History of alcohol abuse at any time in the past;
5. Have received sulfasalazine, azathioprine, 6-mercaptopurine, mycophenolate mofetil, tetracycline, cyclosporine, gold, tacrolimus, sirolimus, or other disease modifying anti-rheumatic drug (DMARD) within 8 weeks of randomization;
6. Use of infliximab, adalimumab, abatacept, certolizumab, golimumab, or tocilizumab within 8 weeks of randomization;
7. Use of leflunomide within 6 months of randomization;
8. Use of etanercept or anakinra within 4 weeks of randomization;
9. Use of a B-cell depleting agent such as rituximab or ocrelizumab, or cytotoxic agents, such as cyclophosphamide or chlorambucil, within one year of randomization;
10. Currently taking cytochrome P450 inhibitors including protease inhibitors such as ritonavir, indinavir, nelfinavir, or macrolide antibiotics such as erythromycin, telithromycin, clarithromycin, or azole antifungals such as fluconazole, ketoconazole, itraconazole, or cimetidine, nefazodone, bergamottin (constituent of grapefruit juice), quercetin, aprepitant, or verapamil;
11. Currently taking cytochrome P450 inducers including St. John's wort, rifampicin, rifabutin, rifapentin, dexamethasone, phenytoin, carbamazapine, phenobarbitol, or troglitazone;
12. Intra-articular, intravenous, or intramuscular corticosteroid injection within 4 weeks of randomization;
13. History or presence of any form of cancer within the 10 years prior to randomization, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
14. Evidence of tuberculosis (TB) based on chest X rays, tuberculin skin test, QuantiFERON®-TB Gold test, or T-SPOT®.
15. Presence of Felty's syndrome, psoriatic arthritis, gout, or other auto-immune diseases;
16. Major surgery (including joint surgery) within 12 weeks prior to randomization;
17. The subject had an infection requiring antibiotic treatment within 4 weeks of randomization;
18. Subject has any evidence of hepatic disease; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), alkaline phosphatase, or bilirubin > 1.5 x the upper limit of normal;
19. Subject has any evidence of renal impairment; serum creatinine > 1.5 x upper limit of normal or estimated Glomerular Filtration Rate (GFR) based on the Cockcroft-Gault equation < 30 mL/min;
20. History or presence of any medical or psychiatric condition or disease, or laboratory abnormality that, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation and may prevent the subject from completing the study
21. Participated in any clinical study of an investigational product including CCX354-C within 30 days or 5 times the half life of the agent, whichever is longer, prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | 12 weeks

SECONDARY OUTCOMES:
The change from baseline to week 12 of Disease Activity Score for 28 Joints using C-reactive proteine (DAS28-CRP) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (41):
- Belgium (3):
  - Brussels
  - Kortrijik
  - Liège
- Czechia (7):
  - Brno
  - Bruntál
  - Hlučín
  - Ostrava-Trebovice
  - Prague
  - Uherské Hradiště
  - Zlín
- Germany (7):
  - Berlin
  - Frankfurt
  - Hanover
  - Herne
  - Leipzig
  - Mainz
  - Würzburg
- Hungary (5):
  - Balatonfüred
  - Békéscsaba
  - Budapest
  - Székesfehérvár
  - Veszprém
- Amsterdam, Netherlands
- Poland (8):
  - Chełm Śląski
  - Elblag
  - Grodzisk Mazowiecki
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
  - Żyrardów
- Romania (7):
  - Bacau
  - Baia Mare
  - Brăila
  - Bucharest
  - Galati
  - Saint Gheorghe, Covasna
  - Târgovişte
- Ukraine (3):
  - Donetsk
  - Kharkiv
  - Kiev